CLINICAL TRIAL: NCT00357188
Title: Open-Label, Multiple Dose Study to Determine the Relative Bioavailability of Atazanavir (ATV) 400 mg Administered With Ritonavir (RTV) and Efavirenz (EFV) Compared to Atazanavir 300 mg Administered With Ritonavir Alone in Healthy Subjects
Brief Title: Dose Finding Confirmation of Atazanavir With Ritonavir and Efavirenz (ATV/RTV + EFV) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-283
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections; Protease Inhibitor
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; efavirenz

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate + Ritonavir
- B (Active Comparator)
  Interventions: Drug: Atazanavir Sulphate + Ritonavir + Efavirenz

INTERVENTIONS:
Drug: Atazanavir Sulphate + Ritonavir — Capsules, Oral, ATV 300 mg + RTV 100 mg, once daily, 10 days.
  Other Names: Reyataz
  Arms: A
Drug: Atazanavir Sulphate + Ritonavir + Efavirenz — Capsules/Tablets, oral, ATV 400 mg + RTV 100 mg + EFV 600 mg, once daily, 14 days.
  Other Names: Reyataz, Sustiva
  Arms: B

SUMMARY:
The purpose of this study is to assess the exposure of Atazanavir 400 mg with Ritonavir 100 mg and with Efavirenz 600 mg compared to Atazanavir 300 mg with 100 mg without Efavirenz in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30
* Men and women who are not of childbearing potential, ages 18-50 years, inclusive

Exclusion Criteria:

* History of seizures or other central nervous system disorders (including migraine headaches)
* history of diagnosed mental illness or suicidal tendencies
* positive screening for Hep B surface antigen
* Hep C antibody
* HIV-1, -2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-07; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To assess the comparability of atazanavir exposure when dosed in the evening as atazanavir 400 mg with ritonavir 100 mg and with efavirenz 600 mg relative to ATV 300 mg and RTV 100 mg alone in healthy subjects

SECONDARY OUTCOMES:
To assess the PK of EFV when coadministered with ATV 400 mg and RTV 100 mg in the evening
To assess the PK of RTV when dosed as ATV 400 mg with RTV 100 mg and with EFV 600 mg in the evening relative to ATV 300 mg with RTV 100 mg alone
To assess the safety and tolerability of ATV and RTV alone and when coadministered with EFV in the evening in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamilton, New Jersey, United States